CLINICAL TRIAL: NCT04345926
Title: Determination of Dose-response Curves Between Propofol Concentration and Intraoperative Electroencephalographic Patterns Until Burst Suppression
Brief Title: Dose-response Curves Between Propofol and Intraoperative Electroencephalographic Patterns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Antonello Penna, Principal Investigator, Anesthesiologist, MD-PhD, University of Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OAIC 938/18
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Propofol Overdose; EEG
Keywords: Propofol; General anesthesia; EEG; Burst suppression
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Dose-response (Experimental): 1. - Concentration of propofol at the loss of consciousness (LOS) will be recorded in the presence of remifentanil (7.5 ng/mL) (LOS time).
  2. - Patients will be intubated and remifentanil will be decreased to 4 ng/mL.
  3. - Concentration of propofol that caused the LOS will be maintained for 20 minutes (Baseline time).
  4. - Propofol will be increased in steps of 0.3 mcg/mL for 7 minutes until an episode of burst suppression will be observed (Burst suppression time).
  EEG activity will be acquired using a SedLine® monitor during the complete protocol.
  Interventions: Drug: Propofol; Device: Electroencephalogram recording

INTERVENTIONS:
Drug: Propofol — Stepped propofol concentration after 20 min of LOS
  Other Names: Dosage increase
Device: Electroencephalogram recording — Acquisition of EEG activity

SUMMARY:
In the world, 230 million surgeries are performed per year and a significant part is performed in patients over 65 years of age. These patients are more labile, especially from the neurocognitive point of view with a high risk to develop neurocognitive complications, such as postoperative delirium. Recent studies have linked this type of complication with an overdose of general anesthetics during surgery. For this reason, in recent years, the use of brain function monitors during the intraoperative period has been recommended to adapt the dosage of the drugs to each patient and thus to avoid overdosing of general anesthetics. However, to date, the available monitors that process the electroencephalographic signal are not able to adequately discriminate gradual changes in anesthetic depth. Also, no systematic studies have been performed that analyze changes that occur in the electroencephalogram (EEG) signal secondary to increases in complications from general anesthetics. Thus, the investigators design this study with the main aim to determine the changes in electroencephalographic patterns induced by a stepped increase of propofol until the burst suppression is reached.

DETAILED DESCRIPTION:
The investigators will carry out a prospective analytical observational clinical study at the Clinical Hospital of the University of Chile. In total 15 patients will be recruited, in who a frontal electroencephalographic signal will be recorded using a SedLine® monitor, and propofol concentration will be estimated using the Marsh model. First, the concentration of propofol at the loss of consciousness (LOS) will be recorded in the presence of remifentanil (7.5 ng/mL). Then, patients will be intubated and remifentanil will be decreased to 4 ng/mL. After that, the concentration of propofol that caused the LOS will be maintained for 20 minutes. Finally, propofol will be increased in steps of 0.3 mcg/mL for 7 min, until an episode of burst suppression will be observed. In the complete protocol, EEG activity will be acquired using a SedLine® monitor.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status 1 or 2
* Low-risk surgery

Exclusion Criteria:

* BMI > 35 kg/m2
* Benzodiazepines use
* Epilepsy
* Psychiatric disorder
* Kidney disease
* Liver disease
* Brain damage

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change in the alpha power of EEG Spectrogram | Change between baseline time (0 minutes) and burst suppression time (35 minutes)
  % of change

SECONDARY OUTCOMES:
Change in the delta power of EEG Spectrogram | Change between baseline time (0 minutes) and burst suppression time (35 minutes)
  % of change
Change in the coherence | Change between baseline time (0 minutes) and burst suppression time (35 minutes)
  % of change
Change in the propofol concentration | Change between baseline time (0 minutes) and burst suppression time (35 minutes)
  concentration in mcg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jose I Egaña, MD/PhD, Principal Investigator — University of Chile; Felipe Maldonado, MD, Principal Investigator — University of Chile; Rodrigo Gutierrez, MD/PhD, Principal Investigator — University of Chile; Antonello Penna, MD/PhD, Principal Investigator — University of Chile
Locations (2):
- Chile (2):
  - Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Hospital Clinico de la Universidad de Chile, Santiago, RM